CLINICAL TRIAL: NCT06747299
Title: The Value of Artificial Intelligence-based 18F-FDG PET/CT in Diferential Diagnosis, Efficacy Prediction and Prognosis Prediction of T-NK Cell Lymphoma: a Clinical Study
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Principal Investigator, GUO RUI, Deputy director, Ruijin Hospital
Other Study IDs: RuijinH 2024-349
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-09

CONDITIONS: T-NK Cell Lymphoma
Keywords: T-NK cell Lymphoma; PET/CT; Diferential Diagnosis; Efficacy Prediction; Prognosis Prediction
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients diagnosis of T-NK cell lymphoma

SUMMARY:
Based on the PET/CT imaging data of patients with T-NK cell lymphoma, machine learning and deep learning methods are used to extract imaging features, establish a T-NK cell lymphoma prediction model, and provide more scientific and accurate prognosis prediction for the clinic.

DETAILED DESCRIPTION:
This study adopts a multicenter retrospective cohort study design，we provided PET/CT of 200 patients with T-NK cell lymphoma as an external validation set for model validation.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological histology confirmed as T-NK Cell Lymphoma; 2.18F-FDG PET/CT examination before treatment; 3. Using modern best practice treatment options; 4. Complete clinicopathological and follow-up data were obtained.

Exclusion Criteria:

1. The patient had previously received antitumor therapy;
2. The patient had a history of other tumors;
3. Incomplete clinical information or imaging data;
4. Concomitant other malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathological histology confirmed as T-NK Cell Lymphoma at Ruijin Hospital, Shanghai JiaoTong University School of Medicine
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation the value of Artificial Intelligence-based 18F-FDG PET/CT of T-NK Cell Lymphoma | Within 1 week of enrollment and after 3 months treatment
  The Value of Artificial Intelligence-based 18F-FDG PET/CT in Diferential Diagnosis, Efficacy Prediction and Prognosis Prediction of T-NK Cell Lymphoma

SECONDARY OUTCOMES:
Progress free survival | 3 years
  Progress free survival
Overall survival | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No